CLINICAL TRIAL: NCT00855218
Title: A Phase II Randomized, Double-blind, Placebo-controlled Study of Sorafenib or Placebo in Combination With Transarterial Chemoembolization (TACE) Performed With DC Bead and Doxorubicin for Intermediate Stage Hepatocellular Carcinoma (HCC).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12918; 2008-005056-24 (EudraCT Number)
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Sorafenib; TACE; DC bead; Combination
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) + TACE (Experimental): Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily). Patients were then also treated with Transarterial Chemoembolization (TACE) performed with DC Bead (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of sorafenib, TACE was also performed on Days 1 (+ 4 days) of cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo + TACE (Placebo Comparator): Placebo was to be orally administered as 2 tablets bid (twice daily). Patients were then also treated with TACE performed with DC Bead (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of placebo, TACE was also performed on Days 1 (+ 4 days) of cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — 800 mg sorafenib (4 tablets) will be taken daily (400mg b.i.d. [twice daily], 2 tablets). Transarterial Chemoembolization (TACE) using DC Bead
  Arms: Sorafenib (Nexavar, BAY43-9006) + TACE
Drug: Placebo — 4 tablets of placebo will be taken daily (2 tablets b.i.d). TACE using DC Bead
  Arms: Placebo + TACE

SUMMARY:
This study will look at whether our drug (sorafenib) in combination with chemotherapy delivered directly into your tumor using beads (DC Bead) will slow the progression of the disease. The beads used with the chemotherapy will slowly release the chemotherapy reducing the adverse effects that normally occur with chemotherapy.

DETAILED DESCRIPTION:
Safety issues will be reported in Adverse Event section. In addition to the secondary outcome measures, Biomarkers and Patient Report Outcome will also be analyzed as other variables.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, multinodular asymptomatic tumor without vascular invasion or extrahepatic spread
* Confirmed Diagnosis of HCC:
* Cirrhotic subjects: Clinical diagnosis by American Association for the Study of Liver Diseases (AASLD) criteria
* HCC can be defined in cirrhotic subjects by one imaging technique (Computed tomography [CT] scan, Magnetic resonance imaging [MRI], or second generation contrast ultrasound) showing a nodule larger than 2 cm with contrast uptake in the arterial phase and washout in venous or late phases or two imaging techniques showing this radiological behavior for nodules of 1-2 cm in diameter.
* Cytohistological confirmation is required for subjects who do not fulfill these eligibility criteria.
* Non-cirrhotic subjects:

For subjects without cirrhosis, histological or cytological confirmation is mandatory

* Documentation of original biopsy for diagnosis is acceptable
* Child Pugh class A without ascites
* Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to randomization:

Exclusion Criteria:

* Patients on a liver transplantation list or with advanced liver disease as defined below:
* Child Pugh B and C
* Active gastrointestinal bleeding
* Encephalopathy
* Ascites
* Lesions having previously been treated with local therapy such as resection of HCC, radiofrequency ablation (RFA), percutaneous ethanol injection (PEI) or cryoablation can not be selected as the target lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (90):
- United States (17):
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Richmond, Virginia
  - Seattle, Washington
- Australia (7):
  - Camperdown, New South Wales
  - St Leonards, New South Wales
  - Greenslopes, Queensland
  - Clayton, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (3):
  - Bruxelles - Brussel
  - Leuven
  - Liège
- Canada (3):
  - Calgary, Alberta
  - Halifax, Nova Scotia
  - Toronto, Ontario
- China (4):
  - Guangzhou, Guangdong
  - Xi'an, Shannxi
  - Beijing
  - Shanghai
- France (7):
  - Créteil
  - Lille
  - Lyon
  - Marseille
  - Paris
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (15):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Erlangen, Bavaria
  - München, Bavaria
  - Regensburg, Bavaria
  - Frankfurt am Main, Hesse
  - Hanover, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Jena, Thuringia
  - Berlin
  - Hamburg
- Italy (10):
  - Bari, Apulia
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Milan, Lombardy
  - Turin, Piedmont
  - Palermo, Sicily
  - Pisa, Tuscany
  - Padua, Veneto
  - Verona, Veneto
- Singapore, Singapore
- South Korea (4):
  - Daegu
  - Gyeonggi-do
  - Seoul
  - Gangnam Severance Hospital, Yonsei University, Seoul
- Spain (15):
  - Santiago de Compostela, A Coruña
  - Badalona, Barcelona
  - Sabadell, Barcelona
  - Cruces/Barakaldo, Bilbao
  - Barcelona, Catalonia
  - Fundación Hospital Alcorcón, Alcorcón, Madrid
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - A Coruña
  - Alicante
  - Barcelona
  - Córdoba
  - Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Valencia
- Taiwan (2):
  - Changhua Christian Hospital, Changhua
  - Taipei

REFERENCES:
- [Derived] Lencioni R, Llovet JM, Han G, Tak WY, Yang J, Guglielmi A, Paik SW, Reig M, Kim DY, Chau GY, Luca A, Del Arbol LR, Leberre MA, Niu W, Nicholson K, Meinhardt G, Bruix J. Sorafenib or placebo plus TACE with doxorubicin-eluting beads for intermediate stage HCC: The SPACE trial. J Hepatol. 2016 May;64(5):1090-1098. doi: 10.1016/j.jhep.2016.01.012. Epub 2016 Jan 22. PMID 26809111
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib (Nexavar, BAY43-9006) + TACE: Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily). Participants were then also treated with Transarterial Chemoembolization (TACE) performed with doxorubicin capable beads (DC Bead) (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of sorafenib, TACE was also performed on Days 1 (+ 4 days) of cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
- Placebo + TACE: Placebo was to be orally administered as 2 tablets bid (twice daily). Participants were then also treated with TACE performed with doxorubicin capable beads (DC Bead) (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of placebo, TACE was also performed on Days 1 (+ 4 days) of cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
Period: Overall Study
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Started | 154 | 153
Participants Received Treatment | 153 | 151
Completed | 0 | 0
Not Completed | 154 | 153
Not completed — Adverse Event | 43 | 27
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Physician Decision | 18 | 11
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 5 | 9
Not completed — non-compliant with study drug | 3 | 1
Not completed — patient convenience | 2 | 0
Not completed — technical problems | 2 | 1
Not completed — Still treated with study medication | 0 | 1
Not completed — Untreatable disease progression | 54 | 67
Not completed — Second malignancy | 0 | 1
Not completed — Progression measurement proven | 7 | 15
Not completed — Clinical endpoint reached | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib (Nexavar, BAY43-9006) + TACE: Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily). Participants were then also treated with Transarterial Chemoembolization (TACE) performed with DC Bead (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of sorafenib, TACE was also performed on Days 1 (+ 4 days) of cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
- Placebo + TACE: Placebo was to be orally administered as 2 tablets bid (twice daily). Participants were then also treated with TACE performed with DC Bead (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of placebo, TACE was also performed on Days 1 (+ 4 days) of cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE | Total
Number analyzed (Participants) | 154 | 153 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (11.9) | 62.7 (11.9) | 62.6 (11.9)
Age, Customized [Number; unit: Participants]
  <65 years | 77 | 82 | 159
  65 - 74 years | 52 | 48 | 100
  >=75 years | 25 | 23 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 135 | 126 | 261
Eastern Cooperative Oncology Group (ECOG) performance status at enrollment [Number; unit: Scores on a scale] — Measures on a scale from grade 0 (best) to grade 5 (worst) cancer's affect on patient's life. 0=Fully active without restriction; 1= Restricted in physically strenuous activity; 2= Ambulatory, capable of all selfcare; 3= Capable of limited selfcare; 4= Completely disabled; 5= Dead
  Scores on a scale
    Missing | 0 | 1 | 1
    Grade 0 | 154 | 152 | 306
Number of target lesions [Number; unit: Participants]
  1 | 30 | 31 | 61
  2 | 58 | 49 | 107
  3 | 33 | 33 | 66
  4 | 12 | 18 | 30
  5 | 21 | 22 | 43
Number of non-target lesions [Number; unit: Participants]
  0 | 72 | 73 | 145
  1 | 40 | 39 | 79
  2 | 24 | 18 | 42
  3 | 7 | 10 | 17
  4 | 3 | 6 | 9
  5 | 4 | 2 | 6
  6 | 0 | 1 | 1
  7 | 1 | 2 | 3
  8 | 1 | 1 | 2
  10 | 1 | 1 | 2
  14 | 1 | 0 | 1
Alfa-fetoprotein [Number; unit: Participants]
  <400 ng/mL | 113 | 112 | 225
  >/=400 ng/mL | 41 | 41 | 82
Child pugh classification [Number; unit: Participants] — Used to assess the severity of a participant's liver disease, the prognosis, and the appropriate treatment. A Child-Pugh class A (well-compensated disease); class B (significant functional compromise); and class C (decompensated disease).
  Participants
    Missing | 0 | 1 | 1
    Class A | 153 | 152 | 305
    Class B | 1 | 0 | 1
Time of first study medication since initial diagnosis [Median (Full Range); unit: Months] — This variable shows time from the first diagnosis of HCC until the first treatment with study drug.
  Months | 1.60 [0.1 to 47.6] | 1.91 [0.1 to 96.4] | 1.71 [0.1 to 96.4]
Time of first study medication since first progression [Median (Full Range); unit: Months] — This variable shows the time from the first treatment with study drug until radiological confirmed disease progression.
  Months | 1.45 [0.2 to 22.0] | 2.56 [0.2 to 28.9] | 1.91 [0.2 to 28.9]
Time of first study medication since most recent progression [Median (Full Range); unit: Months] | 1.02 [0.2 to 6.8] | 1.25 [0.2 to 8.1] | 1.09 [0.2 to 8.1]

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) - Independent Radiological Review (Primary Analysis)
Description: TTP is defined as the time (days) from randomization to radiological confirmed disease progression. Participants without progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: From randomization of the first participant until 28 months later (cut-off date)
Population: Intent-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Number analyzed (Participants) | 154 | 153
Days | 169 [166 to 219] | 166 [113 to 168]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + TACE vs Placebo + TACE; Test type: Superiority or Other; p = 0.072, Log Rank — stratified one-sided (alpha=0.15). adjusted for region and Alfa-fetoprotein (AFP) level at baseline; Hazard Ratio (HR) = 0.797, 95% CI [0.588 to 1.080]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time (days) from randomization to death due to any cause. Participants still alive at the time of analysis were censored at their last date of last contact.
Time Frame: From randomization of the first participant until 28 months later (cut-off date)
Population: Intent-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Number analyzed (Participants) | 154 | 153
Days | NA [554 to NA] — Value cannot be estimated due to censored data | NA [562 to NA] — Value cannot be estimated due to censored data
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + TACE vs Placebo + TACE; Test type: Superiority or Other; p = 0.295, Log Rank; stratified one-sided (alpha=0.15). adjusted for region and AFP level at baseline; Hazard Ratio (HR) = 0.898, 95% CI [0.606 to 1.330]

3. Secondary Outcome: Time to Untreatable Progression (TTUP)
Description: Time to untreatable progression (TTUP) was defined as the time (days) from randomization to untreatable progression. Participants without untreatable progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: From randomization of the first participant until 28 months later (cut-off date)
Population: Intent-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Number analyzed (Participants) | 154 | 153
Days | 95 [62 to 113] | 224 [158 to 288]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + TACE vs Placebo + TACE; Test type: Superiority or Other; p = 0.999, Log Rank; startified one-sided (alpha=0.15), adjusted for region and AFP level at baseline; Hazard Ratio (HR) = 1.586, 95% CI [1.200 to 2.096]

4. Secondary Outcome: Time to Vascular Invasion/Extrahepatic Spread (TTVI/ES)
Description: Time to vascular invasion/extrahepatic spread (TTVI/ES) was defined as the time (days) from randomization to vascular invasion/extrahepatic spread. Participants without vascular invasion/extrahepatic spread at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: From randomization of the first participant until 28 months later (cut-off date)
Population: Intent-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Number analyzed (Participants) | 154 | 153
Days | NA [NA to NA] — Value cannot be estimated due to censored data | NA [NA to NA] — Value cannot be estimated due to censored data
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + TACE vs Placebo + TACE; Test type: Superiority or Other; p = 0.076, Log Rank; stratified one sided (alpha=0.15), adjusted on region and AFP level at baseline; Hazard Ratio (HR) = 0.621, 95% CI [0.321 to 1.200]

5. Secondary Outcome: Tumor Response - Independent Radiological Review
Description: Tumor Response was defined as the number of participants with a confirmed Complete Response (CR)=disappearance of all clinical and radiological tumor lesions, Partial Response (PR)= at least 30% decrease in sum of the longest diameters (LD) of tumor lesions, Stable Disease (SD)= neither sufficient shrinkage to qualify for PR nor sufficient increase for progressive disease, or Progressive Disease (PD)=at least 20% increase in the sum of LD of measured lesions, observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Time Frame: From randomization of the first participant until 28 months later (cut-off date)
Population: Intent-to-treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Number analyzed (Participants) | 154 | 153
Participants
  Response (CR+PR) | 55 | 43
  Complete Response (CR) | 20 | 17
  Partial Response (PR) | 35 | 26
  Stable Disease | 52 | 56
  Progressive Disease | 20 | 36
  Not assessable | 27 | 18

6. Secondary Outcome: Tumor Response - Investigator Assessment
Description: as for outcome 5
Time Frame: From randomization of the first participant until 28 months later (cut-off date)
Population: Intent-to-treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Number analyzed (Participants) | 154 | 153
Participants
  Response (CR+PR) | 66 | 53
  Complete Response | 21 | 20
  Partial Response | 45 | 33
  Stable Disease | 50 | 57
  Progressive Disease | 16 | 30
  Not Assessable | 22 | 13

ADVERSE EVENTS:
Description: Acronyms used: Gastrointestinal (GI), Genitourinary (GU), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Aspartate aminotransferase (AST), Acute respiratory distress syndrome (ARDS), Alanine aminotransferase (ALT), Common Terminology Criteria for Adverse Events (CTCAE)
Groups:
- Sorafenib (Nexavar, BAY43-9006) + TACE: Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily). Patients were then also treated with TACE performed with DC Bead (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of sorafenib on cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
- Placebo + TACE: Placebo was to be orally administered as 2 tablets bid (twice daily). Patients were then also treated with TACE performed with DC Bead (300 to 500 microns) and doxorubicin (150 mg) between 3 to 7 days after the first dose of placebo on cycle 1, 3, 7, 13 and then every 6 cycles thereafter (an optional TACE procedure could be performed between Day 1 of Cycle 7 and Cycle 13 and between Day 1 of Cycles 13 and 19, if deemed necessary by the Investigator.)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + TACE | Placebo + TACE
Serious Adverse Events (participants affected / at risk) | 86/153 | 56/151
Other Adverse Events (participants affected / at risk) | 150/153 | 139/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + TACE (N=153) | Placebo + TACE (N=151)
BLOOD - OTHER (Blood and lymphatic system disorders) | 0 | 1
EDEMA: LIMB (Blood and lymphatic system disorders) | 0 | 1
HEMOGLOBIN (Blood and lymphatic system disorders) | 4 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0
PLATELETS (Blood and lymphatic system disorders) | 1 | 0
CARDIAC GENERAL - OTHER (Cardiac disorders) | 0 | 1
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 3 | 2
CARDIOPULMONARY ARREST (Cardiac disorders) | 1 | 0
HYPERTENSION (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR ARRHYTHMIA, ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
DIABETES (Endocrine disorders) | 2 | 0
ASCITES (Gastrointestinal disorders) | 6 | 2
CONSTIPATION (Gastrointestinal disorders) | 1 | 1
DEHYDRATION (Gastrointestinal disorders) | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GI - OTHER (Gastrointestinal disorders) | 2 | 0
HEARTBURN (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 0 | 1
LEAK, GI, BILIARY TREE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1
PERFORATION, GI, DUODENUM (Gastrointestinal disorders) | 0 | 1
PERFORATION, GI, GALLBLADDER (Gastrointestinal disorders) | 1 | 0
PERFORATION, GI, STOMACH (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 2
CONSTITUTIONAL SYMPTOMS - OTHER (General disorders) | 2 | 0
DEATH NOT ASSOCIATED WITH CTCAE TERM, DISEASE PROGRESSION NOS (General disorders) | 1 | 2
DEATH NOT ASSOCIATED WITH CTCAE TERM, MULTI-ORGAN FAILURE (General disorders) | 0 | 1
DEATH NOT ASSOCIATED WITH CTCAE TERM, SUDDEN DEATH (General disorders) | 0 | 1
FATIGUE (General disorders) | 5 | 1
FEVER (General disorders) | 4 | 6
PAIN, ABDOMEN NOS (General disorders) | 5 | 7
PAIN, BACK (General disorders) | 1 | 0
PAIN, BONE (General disorders) | 1 | 0
PAIN, CHEST WALL (General disorders) | 0 | 1
PAIN, GALLBLADDER (General disorders) | 0 | 1
PAIN, JOINT (General disorders) | 1 | 1
PAIN, PLEURA (General disorders) | 0 | 1
PAIN, STOMACH (General disorders) | 1 | 0
SYNDROMES - OTHER (General disorders) | 2 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 4 | 2
HEPATOBILIARY - OTHER (Hepatobiliary disorders) | 6 | 4
LIVER DYSFUNCTION (Hepatobiliary disorders) | 11 | 5
PANCREATITIS (Hepatobiliary disorders) | 0 | 2
INFECTION (DOCUMENTED CLINICALLY), BLADDER (URINARY) (Infections and infestations) | 1 | 0
INFECTION (DOCUMENTED CLINICALLY), BLOOD (Infections and infestations) | 1 | 2
INFECTION (DOCUMENTED CLINICALLY), BRONCHUS (Infections and infestations) | 0 | 1
INFECTION (DOCUMENTED CLINICALLY), COLON (Infections and infestations) | 0 | 1
INFECTION (DOCUMENTED CLINICALLY), LIVER (Infections and infestations) | 1 | 1
INFECTION (DOCUMENTED CLINICALLY), LUNG (PNEUMONIA) (Infections and infestations) | 3 | 0
INFECTION (DOCUMENTED CLINICALLY), PERITONEAL CAVITY (Infections and infestations) | 2 | 1
INFECTION (DOCUMENTED CLINICALLY), SKIN (CELLULITIS) (Infections and infestations) | 0 | 2
INFECTION (DOCUMENTED CLINICALLY), UPPER AIRWAY NOS (Infections and infestations) | 0 | 1
INFECTION WITH NORMAL ANC, APPENDIX (Infections and infestations) | 1 | 0
INFECTION WITH NORMAL ANC, BILIARY TREE (Infections and infestations) | 1 | 1
INFECTION WITH NORMAL ANC, BLADDER (URINARY) (Infections and infestations) | 0 | 1
INFECTION WITH NORMAL ANC, BLOOD (Infections and infestations) | 4 | 0
INFECTION WITH NORMAL ANC, LIVER (Infections and infestations) | 1 | 0
INFECTION WITH NORMAL ANC, PERITONEAL CAVITY (Infections and infestations) | 1 | 1
INFECTION WITH NORMAL ANC, SKIN (CELLULITIS) (Infections and infestations) | 1 | 0
INFECTION WITH NORMAL ANC, URINARY TRACT NOS (Infections and infestations) | 0 | 1
INFECTION WITH UNKNOWN ANC, BONE (OSTEOMYELITIS) (Infections and infestations) | 1 | 0
INFECTION WITH UNKNOWN ANC, LUNG (PNEUMONIA) (Infections and infestations) | 2 | 1
INFECTION WITH UNKNOWN ANC, PANCREAS (Infections and infestations) | 0 | 1
ALKALINE PHOSPHATASE (Metabolism and nutrition disorders) | 1 | 0
ALT (Metabolism and nutrition disorders) | 6 | 0
AMYLASE (Metabolism and nutrition disorders) | 1 | 0
AST (Metabolism and nutrition disorders) | 7 | 0
BILIRUBIN (HYPERBILIRUBINEMIA) (Metabolism and nutrition disorders) | 5 | 1
CREATININE (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0
LIPASE (Metabolism and nutrition disorders) | 2 | 2
METABOLIC/LAB - OTHER (Metabolism and nutrition disorders) | 0 | 1
FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 2
JOINT-FUNCTION (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE WEAKNESS, LEFT-SIDED (Musculoskeletal and connective tissue disorders) | 0 | 1
SECONDARY MALIGNANCY (POSSIBLY RELATED TO CANCER TREATMENT) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 | 0
CONFUSION (Nervous system disorders) | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 6 | 1
SEIZURE (Nervous system disorders) | 1 | 0
OBSTRUCTION, GU, PROSTATE (Renal and urinary disorders) | 0 | 1
RENAL - OTHER (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 3
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 | 0
ULCERATION (Skin and subcutaneous tissue disorders) | 0 | 1
ARTERY INJURY, EXTREMITY - LOWER (Vascular disorders) | 1 | 1
ARTERY INJURY, OTHER NOS (Vascular disorders) | 1 | 0
HEMORRHAGE PULMONARY, BRONCHOPULMONARY NOS (Vascular disorders) | 1 | 0
HEMORRHAGE WITH SURGERY (Vascular disorders) | 1 | 1
HEMORRHAGE, GI, ABDOMEN NOS (Vascular disorders) | 2 | 1
HEMORRHAGE, GI, ESOPHAGUS (Vascular disorders) | 1 | 0
HEMORRHAGE, GI, LIVER (Vascular disorders) | 1 | 0
HEMORRHAGE, GI, LOWER GI NOS (Vascular disorders) | 2 | 0
HEMORRHAGE, GI, PERITONEAL CAVITY (Vascular disorders) | 0 | 2
HEMORRHAGE, GI, RECTUM (Vascular disorders) | 1 | 0
HEMORRHAGE, GI, STOMACH (Vascular disorders) | 3 | 1
HEMORRHAGE, GI, UPPER GI NOS (Vascular disorders) | 1 | 2
HEMORRHAGE, GI, VARICES (ESOPHAGEAL) (Vascular disorders) | 3 | 4
HEMORRHAGE, GI, VARICES (RECTAL) (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL ISCHEMIA (Vascular disorders) | 1 | 0
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 | 0
VASCULAR - OTHER (Vascular disorders) | 1 | 0
VISCERAL ARTERIAL ISCHEMIA (Vascular disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + TACE (N=153) | Placebo + TACE (N=151)
EDEMA: LIMB (Blood and lymphatic system disorders) | 7 | 16
HEMOGLOBIN (Blood and lymphatic system disorders) | 13 | 9
PLATELETS (Blood and lymphatic system disorders) | 16 | 3
HYPERTENSION (Cardiac disorders) | 46 | 27
DIABETES (Endocrine disorders) | 0 | 8
ANOREXIA (Gastrointestinal disorders) | 48 | 31
ASCITES (Gastrointestinal disorders) | 25 | 22
CONSTIPATION (Gastrointestinal disorders) | 29 | 27
DIARRHEA (Gastrointestinal disorders) | 81 | 28
DISTENSION (Gastrointestinal disorders) | 10 | 11
GASTRITIS (Gastrointestinal disorders) | 10 | 7
GI - OTHER (Gastrointestinal disorders) | 16 | 13
HEARTBURN (Gastrointestinal disorders) | 5 | 10
MUCOSITIS (FUNCTIONAL/SYMPTOMATIC), ORAL CAVITY (Gastrointestinal disorders) | 16 | 6
NAUSEA (Gastrointestinal disorders) | 59 | 58
VOMITING (Gastrointestinal disorders) | 27 | 40
FATIGUE (General disorders) | 65 | 50
FEVER (General disorders) | 56 | 49
FLU-LIKE SYNDROME (General disorders) | 6 | 12
INSOMNIA (General disorders) | 19 | 23
PAIN, ABDOMEN NOS (General disorders) | 93 | 91
PAIN, BACK (General disorders) | 12 | 14
PAIN, CHEST/THORAX NOS (General disorders) | 9 | 6
PAIN, EXTREMITY-LIMB (General disorders) | 6 | 8
PAIN, HEAD/HEADACHE (General disorders) | 13 | 6
PAIN, JOINT (General disorders) | 13 | 15
PAIN, LIVER (General disorders) | 6 | 11
PAIN, MUSCLE (General disorders) | 18 | 11
PAIN, STOMACH (General disorders) | 7 | 11
RIGORS/CHILLS (General disorders) | 11 | 6
WEIGHT LOSS (General disorders) | 31 | 16
ALT (Metabolism and nutrition disorders) | 22 | 25
AMYLASE (Metabolism and nutrition disorders) | 8 | 9
AST (Metabolism and nutrition disorders) | 34 | 29
BILIRUBIN (HYPERBILIRUBINEMIA) (Metabolism and nutrition disorders) | 21 | 13
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 8 | 15
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 19 | 10
HYPOKALEMIA (Metabolism and nutrition disorders) | 16 | 4
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 8 | 2
LIPASE (Metabolism and nutrition disorders) | 18 | 12
METABOLIC/LAB - OTHER (Metabolism and nutrition disorders) | 8 | 6
DIZZINESS (Nervous system disorders) | 12 | 5
MOOD ALTERATION, ANXIETY (Nervous system disorders) | 8 | 12
URINARY FREQUENCY (Renal and urinary disorders) | 8 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 13
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 13 | 8
VOICE CHANGES (Respiratory, thoracic and mediastinal disorders) | 9 | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 43 | 11
DERMATOLOGY - OTHER (Skin and subcutaneous tissue disorders) | 11 | 7
DRY SKIN (Skin and subcutaneous tissue disorders) | 16 | 6
HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 71 | 10
PRURITUS (Skin and subcutaneous tissue disorders) | 13 | 18
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 33 | 11
HEMORRHAGE PULMONARY, NOSE (Vascular disorders) | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must discuss and obtain written consent of the sponsor on the intended publication. The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of the submission inorder to obtain approval.